CLINICAL TRIAL: NCT05294328
Title: A Multicenter, Double-Masked Evaluation of the Safety and Effectiveness of Aceclidine /Brimonidine (LNZ101) and Aceclidine (LNZ100) in the Treatment of Presbyopia
Brief Title: Evaluation of the Safety and Effectiveness of Aceclidine/Brimonidine (LNZ101) and Aceclidine (LNZ100) in the Treatment of Presbyopia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LENZ Therapeutics, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-100-0007
Record Dates: First submitted 2022-03-04; First posted 2022-03-24 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Presbyopia; Refractive Errors; Eye Diseases
Keywords: Pharmaceutical Solutions; Miotics; Ophthalmic Solutions; Near Vision; Eye Drops; INSIGHT 1
MeSH Terms: conditions — Presbyopia; Refractive Errors; Eye Diseases; Myopia | interventions — Brimonidine Tartrate; aceclidine

STUDY DESIGN:
Intervention Model Description: Multicenter, double-masked, randomized, crossover, active and vehicle-controlled, safety and effectiveness study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Combination ophthalmic solution (LNZ101) dosed bilaterally (Experimental): LNZ101: Aceclidine/Brimonidine combination ophthalmic solution
  Interventions: Drug: Aceclidine+Brimonidine combination ophthalmic solution
- Aceclidine Ophthalmic Solution (LNZ100) dosed bilaterally (Experimental): LNZ100: Aceclidine ophthalmic solution
  Interventions: Drug: Aceclidine ophthalmic solution
- Vehicle Ophthalmic Solution dosed bilaterally (Experimental): Proprietary Vehicle ophthalmic solution
  Interventions: Drug: Vehicle Proprietary Ophthalmic Solution

INTERVENTIONS:
Drug: Aceclidine+Brimonidine combination ophthalmic solution — LNZ101-combination ophthalmic solution
  Other Names: LNZ101; Brimonidine and Aceclidine
  Arms: Combination ophthalmic solution (LNZ101) dosed bilaterally
Drug: Aceclidine ophthalmic solution — LNZ100- aceclidine ophthalmic solution
  Other Names: LNZ100; Aceclidine
  Arms: Aceclidine Ophthalmic Solution (LNZ100) dosed bilaterally
Drug: Vehicle Proprietary Ophthalmic Solution — Proprietary Vehicle Ophthalmic Solution
  Other Names: Vehicle
  Arms: Vehicle Ophthalmic Solution dosed bilaterally

SUMMARY:
To evaluate the safety and effectiveness of Aceclidine/Brimonidine (LNZ101) compared with Aceclidine (LNZ100) and vehicle in the treatment of Presbyopia.

ELIGIBILITY:
Inclusion Criteria:

Subjects MUST:

1. Be able and willing to provide written informed consent and sign Health Information Portability and Accountability Act (HIPAA) form prior to any study procedure being performed;
2. Be able and willing to follow all instructions and attend study visits;
3. Be 45-75 years of age of either sex and any race or ethnicity at Visit 1;
4. Have +1.00 to -4.00 diopter (D) of sphere (so that SE results in myopia no more severe than -4.00 SE. See Inclusion 5 below) in both eyes determined by manifest refraction documented at Visit 1;
5. Have up to 2.00D of cylinder (minus cylinder) in both eyes determined by manifest refraction documented at Visit 1;
6. Be presbyopic as determined at Visit 1

Exclusion Criteria:

Subjects must NOT:

1. Be a female of childbearing potential who is currently pregnant, nursing or planning a pregnancy;
2. Have known contraindications or sensitivity to the use of any of the study medications(s) or their components;
3. Have an active ocular infection at Visit 1 (bacterial, viral or fungal), positive history of an ocular herpetic infection, preauricular lymphadenopathy, or ongoing, active ocular inflammation (e.g., moderate to severe blepharitis, allergic conjunctivitis, peripheral ulcerative keratitis, scleritis, uveitis) in either eye;
4. Have moderate or severe dry eye determined by total corneal fluorescein staining at Visit 1;
5. Have clinically significant abnormal lens findings (e.g., cataract) including early lens changes and/or any evidence of a media opacity in either eye during dilated slit-lamp biomicroscopy and fundus exam documented within 3 months of Visit 1;

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alisyn Facemire, BA, Study Director — LENZ Therapeutics, Inc
Locations (5):
- United States (5):
  - INSIGHT-1 Study Site #4, Glendale, California
  - INSIGHT-1 Study Site #3, Indianapolis, Indiana
  - INSIGHT-1 Study Site #1, Andover, Massachusetts
  - INSIGHT-1 Study Site #2, Memphis, Tennessee
  - INSIGHT-1 Study Site #5, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Crossover Sequence 1 (123): LNZ101 (1), LNZ100 (2), Vehicle (3)
- Crossover Sequence 2 (231): LNZ100 (2), Vehicle (3), LNZ101 (1)
- Crossover Sequence 3 (312): Vehicle (3), LNZ101 (1), LNZ100 (2)
Period: Overall Study
Arm/Group | Crossover Sequence 1 (123) | Crossover Sequence 2 (231) | Crossover Sequence 3 (312)
Started | 22 | 22 | 24
Completed | 20 | 18 | 23
Not Completed | 2 | 4 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Other (Corneal Surface Disease and Distance VA) | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crossover Sequence 1 (123) | Crossover Sequence 2 (231) | Crossover Sequence 3 (312) | Total
Number analyzed (Participants) | 22 | 22 | 24 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (6.37) | 55.7 (6.02) | 55.5 (6.04) | 56.2 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 10 | 41
  Male | 6 | 7 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 7 | 18
  Not Hispanic or Latino | 17 | 16 | 17 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 5 | 10
  White | 18 | 16 | 19 | 53
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥ 3-line Improvement in Near Vision and no Loss ≥ 5 Letters Distance Vision
Description: Percentage of participants with at least a 3-line improvement in near vision and no loss ≥ 5 letters distance vision
Time Frame: 1 hour post treatment
Population: The treatment crossover design allowed for each treatment to be analyzed in all subjects. The primary efficacy analysis was performed on a mITT population of subjects meeting the baseline criteria.
Measure: Number; unit: percentage of participants
Groups:
- LNZ101: LNZ101 (aceclidine hydrochloride and brimonidine tartrate) (non-preserved) Ophthalmic Solution
- LNZ100: LNZ100 (Aceclidine hydrochloride) (non-preserved) Ophthalmic solution
- Vehicle Ophthalmic Solution: Vehicle Proprietary Ophthalmic Solution
Arm/Group | LNZ101 | LNZ100 | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 50 | 49 | 51
percentage of participants | 56.0 | 71.4 | 5.9
Statistical Analysis 1: Comparison: LNZ101 vs Vehicle Ophthalmic Solution; Test type: Superiority; p < 0.0001, Generalized Estimating Equation (GEE); Odds Ratio (OR) = 34.262
Statistical Analysis 2: Comparison: LNZ100 vs Vehicle Ophthalmic Solution; Test type: Superiority; p < 0.0001, Generalized Estimating Equation (GEE); Odds Ratio (OR) = 73.443

ADVERSE EVENTS:
Time Frame: Approximately 3 weeks
Groups:
- Vehicle Ophthalmic Solution: Proprietary Vehicle ophthalmic solution
Arm/Group | LNZ101 | LNZ100 | Vehicle Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62 | 0/61
Other Adverse Events (participants affected / at risk) | 9/62 | 3/62 | 8/61
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LNZ101 (N=62) | LNZ100 (N=62) | Vehicle Ophthalmic Solution (N=61)
Ocular Vision Blurred (Eye disorders) | 0 | 0 | 7
Non-Ocular Headache (Nervous system disorders) | 9 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT05294328/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT05294328/SAP_001.pdf